CLINICAL TRIAL: NCT01318083
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of SYR-322 When Used in Combination With Sulfonylurea in Subjects With Type 2 Diabetes in Japan
Brief Title: Efficacy and Safety of Alogliptin Used in Combination With Sulfonylurea in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322/CCT-005; UMIN000001393 (Registry Identifier: UMIN-CTR); JapicCTI-080626 (Registry Identifier: JapicCTI); U1111-1119-6261 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD and Glimepiride QD or BID (Active Comparator)
  Interventions: Drug: Alogliptin and glimepiride
- Alogliptin 25 mg QD and Glimepiride QD or BID (Active Comparator)
  Interventions: Drug: Alogliptin and glimepiride
- Glimepiride 1, 2, 3 or 4 mg QD or BID (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Alogliptin and glimepiride — Alogliptin 12.5 mg, tablets, orally, once daily and glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily for up 12 weeks.
  Other Names: SYR-322; Amaryl
  Arms: Alogliptin 12.5 mg QD and Glimepiride QD or BID
Drug: Alogliptin and glimepiride — Alogliptin 25 mg, tablets, orally, once daily and glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily for up 12 weeks.
  Other Names: SYR-322; Amaryl
  Arms: Alogliptin 25 mg QD and Glimepiride QD or BID
Drug: Glimepiride — Glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily and alogliptin placebo-matching tablets, orally, once daily for up 12 weeks.
  Other Names: Amaryl
  Arms: Glimepiride 1, 2, 3 or 4 mg QD or BID

SUMMARY:
The purpose of this study was evaluate the efficacy and safety of alogliptin, once daily (QD) combined with an Sulfonylurea taken QD or twice daily (BID) in type 2 diabetic patients with uncontrolled blood glucose.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

The present study was planned to evaluate the efficacy and safety of alogliptin as an add-on to sulfonylurea in type 2 diabetic patients who had uncontrolled blood glucose despite treatment with an sulfonylurea as well as diet and exercise therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Had been taking a sulfonylurea for at least 4 weeks prior to the initiation of the observation period (Week -12).
2. Had been taking glimepiride at a stable dose regimen (1, 2, 3 or 4 mg/day, once or twice daily in the morning or in the morning and evening, before or after meal) for at least 12 weeks prior to the initiation of the treatment period (Week 0).
3. Had glycosylated hemoglobin (HbA1c) of 7.0% or more and below 10.0% at 8 weeks after the initiation of the observation period (Week -4).
4. Had an HbA1c difference between 4 weeks after the initiation of the observation period (Week -8) and 8 weeks after the initiation of the observation period (Week -4) being within 10.0%* of the value at 4 weeks after the initiation of the observation period (Week -8) (*rounded off to the first decimal place).
5. Was receiving specific diet and exercise (if any) therapies during the observation period.

Exclusion Criteria:

1. Had taken other diabetic medications than glimepiride within 12 weeks before the initiation of the treatment period (Week 0).

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Professor, Diabetes and Endocrine Division, Study Director — Department of Medicine, Kawasaki Medical School

REFERENCES:
- [Derived] Seino Y, Hiroi S, Hirayama M, Kaku K. Efficacy and safety of alogliptin added to sulfonylurea in Japanese patients with type 2 diabetes: A randomized, double-blind, placebo-controlled trial with an open-label, long-term extension study. J Diabetes Investig. 2012 Dec 20;3(6):517-25. doi: 10.1111/j.2040-1124.2012.00226.x. Epub 2012 Jul 12. PMID 24843617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 33 investigative sites in Japan from 20 August 2008 to 18 April 2009.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with uncontrolled blood glucose despite treatment with sulfonylurea as well as diet and exercise therapies were enrolled in one of 3, once-daily (QD) or twice daily (BID) treatment groups.
Groups:
- Alogliptin 12.5 mg QD and Glimepiride QD or BID: Alogliptin 12.5 mg, tablets, orally, once daily and glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily for up 12 weeks.
- Alogliptin 25 mg QD and Glimepiride QD or BID: Alogliptin 25 mg, tablets, orally, once daily and glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily for up 12 weeks.
- Glimepiride 1, 2, 3 or 4 mg QD or BID: Glimepiride 1, 2, 3 or 4 mg, tablets, orally, once or twice daily and alogliptin placebo-matching tablets, orally, once daily for up 12 weeks.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Started | 105 | 104 | 103
Completed | 99 | 102 | 98
Not Completed | 6 | 2 | 5
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Treatment Complications | 1 | 0 | 0
Not completed — Lack of Study Medication Compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID | Total
Number analyzed (Participants) | 105 | 104 | 103 | 312
Age, Customized [Number; unit: participants]
  ≤ 64 years | 66 | 73 | 64 | 203
  ≥ 65 years | 39 | 31 | 39 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 32 | 108
  Male | 66 | 67 | 71 | 204

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Analysis based on last observation carried forward, where the last postbaseline double-blind observed value is carried forward and used for all subsequent scheduled time points where data is missing. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
percentage of Glycosylated Hemoglobin | -0.60 (0.563) | -0.66 (0.564) | 0.34 (0.611)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.936, 95% CI 2-sided [-1.097 to -0.775]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.998, 95% CI 2-sided [-1.160 to -0.837]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 2).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
percentage of Glycosylated Hemoglobin | -0.12 (0.244) | -0.13 (0.206) | 0.08 (0.229)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.196, 95% CI 2-sided [-0.261 to -0.131]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.213, 95% CI 2-sided [-0.273 to -0.154]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
percentage of Glycosylated Hemoglobin | -0.32 (0.357) | -0.36 (0.339) | 0.09 (0.351)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.410, 95% CI 2-sided [-0.507 to -0.312]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.453, 95% CI 2-sided [-0.547 to -0.358]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
percentage of Glycosylated Hemoglobin | -0.52 (0.488) | -0.59 (0.504) | 0.18 (0.525)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.695, 95% CI 2-sided [-0.834 to -0.556]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.770, 95% CI 2-sided [-0.911 to -0.629]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
mg/dL | -17.5 (26.05) | -17.4 (29.19) | 0.2 (24.12)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -17.71, 95% CI 2-sided [-24.60 to -10.83]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -17.59, 95% CI 2-sided [-24.93 to -10.25]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
mg/dL | -21.2 (27.33) | -22.9 (29.33) | 2.0 (24.83)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -23.17, 95% CI 2-sided [-30.33 to -16.02]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -24.88, 95% CI 2-sided [-32.33 to -17.43]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
mg/dL | -22.3 (26.40) | -17.4 (28.88) | 5.3 (29.75)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -27.62, 95% CI 2-sided [-35.32 to -19.91]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -22.72, 95% CI 2-sided [-30.76 to -14.69]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 or final visit and baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 104 | 104 | 103
mg/dL | -22.3 (31.05) | -15.9 (28.12) | 6.0 (32.97)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -28.37, 95% CI 2-sided [-37.14 to -19.59]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -21.93, 95% CI 2-sided [-30.33 to -13.54]

9. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 12).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 12 or final visit and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Number analyzed (Participants) | 101 | 103 | 99
mg/dL | 76.6 (41.51) | 80.9 (50.08) | 100.0 (52.44)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -23.41, 95% CI 2-sided [-36.58 to -10.23]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD and Glimepiride QD or BID vs Glimepiride 1, 2, 3 or 4 mg QD or BID; Test type: Superiority or Other; Mean Difference (Final Values) = -19.18, 95% CI 2-sided [-33.40 to -4.95]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride QD or BID | Alogliptin 25 mg QD and Glimepiride QD or BID | Glimepiride 1, 2, 3 or 4 mg QD or BID
Serious Adverse Events (participants affected / at risk) | 3/105 | 1/104 | 0/103
Other Adverse Events (participants affected / at risk) | 27/105 | 40/104 | 36/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Glimepiride QD or BID (N=105) | Alogliptin 25 mg QD and Glimepiride QD or BID (N=104) | Glimepiride 1, 2, 3 or 4 mg QD or BID (N=103)
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Glimepiride QD or BID (N=105) | Alogliptin 25 mg QD and Glimepiride QD or BID (N=104) | Glimepiride 1, 2, 3 or 4 mg QD or BID (N=103)
Nasopharyngitis (Infections and infestations) | 20 | 20 | 22
Headache (Nervous system disorders) | 0 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 4
Gastroenteritis (Infections and infestations) | 4 | 0 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.